CLINICAL TRIAL: NCT07275333
Title: Human Papillomavirus Self-sampling for Enhancing Cervical Screening During the War in Ukraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Union for International Cancer Control (Other); Zaporizhzhiya State Medical University (Other); World Against Cancer Foundation (Other)
Responsible Party: Principal Investigator, Sara Arroyo Mühr, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-06579-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer; Cervical Cancer Screening; Human Papillomavirus (HPV) Infection; Cervical Intraepithelial Neoplasia
Keywords: hpv self-sampling; hpv testing; cervical cancer prevention; cervical screening; implementation science; war-affected regions; ukraine; High-risk HPV; self-collection; Screening uptake
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Infections; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention consisting of HPV self-sampling and HPV DNA testing. There is no control or comparator arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV Self-Sampling for Cervical Cancer Screening (Experimental): Participants will receive an HPV self-sampling kit distributed through primary care providers, community outreach, or partner organizations in conflict-affected areas of southeastern Ukraine. Women will collect a vaginal sample using the supplied FLOQSwab® device. Samples will be tested for high-risk HPV in quality-assured Ukrainian molecular laboratories. Results will be reported through the project's secure digital platform, which will coordinate follow-up care for HPV-positive women according to clinical guidelines. All participants in this arm receive the same screening intervention.
  Interventions: Device: HPV Self-Sampling Kit

INTERVENTIONS:
Device: HPV Self-Sampling Kit — Participants will receive an HPV self-sampling kit consisting of a sterile vaginal swab and collection tube for home or clinic-based sample collection. The kit includes illustrated instructions to enable unsupervised self-sampling. Women collect the sample themselves and return it. Samples are tested for high-risk HPV using validated PCR-based assays in Ukrainian molecular laboratories participating in the project. Results are communicated through a secure digital platform, which coordinates appropriate clinical follow-up for HPV-positive women. All enrolled participants receive the same intervention.
  Other Names: FLOQSwab® self-collection device; self-sampling

SUMMARY:
In 2020, a cervical screening center was established in Zaporizhzhia (Ukraine), initiating a pilot project to evaluate the prevalence of HPV among women in Eastern Ukraine. The findings were intended to lay the groundwork for the Ukrainian Ministry of Health in establishing a structured national screening program. However, all efforts were halted due to the nearby armed conflict, situated just 40 kilometers from the border.

The World Health Organization's goal to eliminate cervical cancer globally has a gap when it comes to managing cancer control during crises like armed conflicts. We propose a demonstration project to assess whether a simpler, yet modern, cervical cancer control strategy (based on using self-sampling for HPV detection) could also be effective for cervical cancer screening in Zaporizhzhia.

Women aged 30-60 years who have not had a recent negative HPV test will be invited to participate. Participants receive a self-sampling kit from their primary care provider and can return the sample free of charge to the clinic or community volunteers. All samples are analyzed in accredited laboratories in Zaporizhzhia.

HPV-positive women will receive follow-up care according to national guidelines, including referral to gynecologists for additional tests and treatment if needed. HPV-negative women will be reassured and advised on future screening intervals.

The study also evaluates how well the screening program can be implemented during conflict conditions. This includes measuring women's acceptance of self-sampling, the willingness of providers to adopt the procedures, and whether the screening process is feasible, practical, and sustainable. Additional process evaluation will explore how the program adapts to challenges such as migration, disrupted health services, and safety concerns.

This project is conducted through collaboration between Zaporizhzhia State Medical and Pharmaceutical University, the Charitable Foundation "World Against Cancer," and Karolinska Institutet in Sweden, which provides quality assurance support for laboratory procedures. The goal is to establish a safe, effective, and sustainable cervical cancer screening model that can be used in conflict-affected regions and similar settings.

This work is supported by a grant from the Union for International Cancer Control (UICC), as part of the Reimagining Cancer Research in Europe Initiative.

DETAILED DESCRIPTION:
Cervical cancer is the fourth leading cause of cancer-related deaths among women worldwide and is almost always caused by persistent infection with high-risk human papillomavirus (HPV). Organized screening programs using HPV testing have been shown to reduce cervical cancer incidence and mortality. However, in settings affected by armed conflict, access to preventive services is disrupted, and clinic-based screening becomes difficult to maintain.

In 2020, a cervical screening center was established in the Zaporizhzhia region of Ukraine, close to the conflict zone. A pilot HPV-based screening initiative was launched to estimate HPV prevalence and support the development of an organized national screening program. This effort was interrupted by the escalation of the war, which led to disruption of services, population displacement, and increased barriers to preventive care.

This study aims to revive and expand these efforts by implementing an HPV-based cervical cancer screening program using self-sampling in Zaporizhzhia. The project leverages the long-standing experience from Sweden in organized screening, HPV laboratory quality assurance, and self-sampling implementation, while adapting the model to conflict-affected conditions in Ukraine.

Objectives

The main objectives are to:

* Improve access to cervical cancer screening for women in Zaporizhzhia by offering HPV testing on self-collected samples.
* Ensure accurate and reliable HPV testing through participation in external proficiency schemes and the use of accredited laboratories.
* Provide timely and guideline-based follow-up for women who test positive for high-risk HPV.
* Evaluate key implementation outcomes (e.g., acceptability, adoption, appropriateness, feasibility).
* Conduct a process evaluation to understand how the intervention is adapted and sustained in the context of ongoing conflict.

Study Design and Intervention

Women aged 30-60 years living in Zaporizhzhia who have not had a documented negative HPV test in the past three years will be eligible. No exclusions are made based on socioeconomic status or ethnicity. Women with prior hysterectomy or inability to provide informed consent will be excluded.

The intervention comprises several coordinated components:

1. Quality assurance of HPV testing:

   Two PCR laboratories in Zaporizhzhia participate in annual external proficiency testing coordinated by the International HPV Reference Center. One laboratory serves as the primary testing site and a second as a contingency laboratory. Only assays that achieve proficiency for high-risk HPV detection will be used.
2. Centralized database:

   A secure electronic platform (selfsamplingukraine.ua) is developed to collect/register: patient registration, risk classification, kit distribution, patient feedback and HPV test results. The database functions both as a clinical registry and as the primary data source for monitoring, evaluation, and implementation outcomes.
3. Protocols and training:

   Standard operating procedures define eligibility criteria, self-sampling instructions, sample handling, HPV testing, result reporting, and follow-up pathways. Healthcare providers receive structured training on these procedures, including how to counsel women, interpret HPV results, and arrange follow-up.
4. Self-sampling and HPV testing:

   Primary care physicians and collaborating partners (NGOs) distribute self-sampling kits with written instructions. Women can return the samples directly to clinics, or via volunteers from the Charitable Foundation "World Against Cancer." Collected samples are tested for high-risk HPV types in the accredited laboratories. Regular internal and external quality controls are performed.
5. Result reporting and follow-up:

   HPV test results are uploaded to the secure platform and made available to the woman's primary care physician, who then informs the participant and organises follow-up. Women with HPV 16/18 are prioritised for expedited gynaecological assessment (colposcopy) within two months. Women with other high-risk HPV types are managed according to national or project-specific guidelines (e.g., repeat testing at 12 months or referral for colposcopy). HPV-negative women are reassured and advised on routine screening intervals.
6. Implementation and Process Evaluation

An embedded implementation research and process evaluation component will assess how the intervention functions in a conflict-affected setting. Data sources include: a) Routine registry data participation, kit return rates, HPV positivity, and follow-up completion; b) Structured surveys of participants to measure acceptability, perceived barriers and facilitators, and satisfaction with self-sampling and follow-up; c) Surveys and semi-structured interviews with healthcare providers and key stakeholders to assess adoption, appropriateness, feasibility, workload, and perceived sustainability; d) review of project documents, meeting minutes, and timelines to document adaptations over time.

Quantitative analyses will use descriptive statistics for participation and HPV outcomes and, where relevant, comparative analyses to explore factors associated with screening uptake and follow-up completion. Qualitative data will be analysed thematically to identify key themes regarding acceptability, feasibility, and contextual influences.

Target Population and Expected Impact

The anticipated sample size is approximately 1,000 women, corresponding to the estimated number of eligible women reachable within the current healthcare system in Zaporizhzhia. All eligible women who consent will be included.

The target population is women aged 30-60 years living in Zaporizhzhia, a region affected by war and health system disruption. The intervention is expected to:

* Increase access to screening by offering a convenient self-sampling option.
* Enable earlier detection of high-risk HPV infections and precancerous lesions.
* Reduce the burden of advanced cervical cancer and the associated physical, emotional, and economic consequences.
* Provide an evidence-based, scalable model for cervical cancer screening in conflict and other resource-constrained settings.

The study also aims to reduce inequalities in access to preventive services by prioritising outreach and free participation for women who might otherwise be missed by traditional clinic-based screening.

Ethical Approval

Ethical approval has been granted by the Ethics Committee of the Educational and Scientific Medical Center "University Clinic," Zaporizhzhia State Medical and Pharmaceutical University (Protocol No. 9, 24 September 2024, with earlier approvals). Karolinska Institutet has received approval from the Swedish Ethical Review Authority (2024-06579-01) to conduct quality assurance activities related to the project.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 30-60 years
* Intact uterus (no prior hysterectomy)
* Eligible for cervical cancer screening according to local guidelines
* Able to provide informed consent
* Able to perform self-sampling at home or at a clinic

Exclusion Criteria:

* History of total hysterectomy
* Pregnancy at the time of enrollment
* Known diagnosis of cervical cancer
* Inability or unwillingness to provide informed consent
* Unable to perform self-sampling or comply with study procedures

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of HPV self-sampling among eligible women in Zaporizhzhia | Up to 12 weeks after receipt of the self-sampling kit.
  Proportion of eligible women aged 30-60 who receive an HPV self-sampling kit and return a valid sample for testing. This outcome reflects the feasibility and adoption of the screening intervention during wartime conditions and directly corresponds to the project objective of improving access to cervical cancer screening through self-sampling.

SECONDARY OUTCOMES:
Acceptability of HPV self-sampling among participants | Within 4 weeks after sample return
  Participant acceptability measured through brief surveys and semi-structured interviews assessing comfort, ease of use, clarity of instructions, and overall satisfaction with self-sampling and follow-up procedures. Designed to evaluate acceptability according to implementation science outcomes.
Adoption of the screening intervention by healthcare providers | Up to 3 months after provider training.
  Number and proportion of primary care providers trained who offer self-sampling, register participants in the database, and report results. Includes qualitative feedback on provider experience, appropriateness, and barriers to implementation as described in the project plan.
Feasibility of implementing HPV self-sampling during conflict | At 12 months and at project completion (up to 24 months post-initiation).
  Assessment of logistical feasibility including kit distribution pathways, sample return methods (post, clinic, NGO volunteers), laboratory capacity, screening workflow continuity, and challenges related to resource availability or security conditions. Based directly on feasibility indicators in the UICC proposal.
Proportion of women who have never been screened prior to participation | At enrollment
  Percentage of enrolled women who report no prior cervical cancer screening or no HPV test within the past 3 years. This evaluates reach and equity of the intervention, as outlined in the project's objectives.
Performance and reliability of locally used HPV tests | At annual proficiency testing cycles (0,12,18 months) and at each HPV test run (up to 24 months).
  Proportion of valid HPV test results and laboratory concordance based on internal quality checks and participation in the International HPV Reference Center proficiency program. This aligns with the quality assurance aims in the UICC plan.
Functionality and use of the digital screening platform | At 6, 12, 18, and 24 months after platform deployment.
  Evaluation of the centralized database (selfsamplingukraine.ua), including completeness of entries, timeliness of result reporting, and usability by providers and participants. Links directly to objectives on data management and monitoring.
Follow-up completion among HPV-positive women | Within 2 months of a positive HPV result.
  Proportion of HPV-positive women who complete recommended follow-up (e.g., referral to gynecologist, colposcopy, repeat HPV testing after 12 months). Reflects fidelity to follow-up protocols defined in the project plan.

CONTACTS AND LOCATIONS:
Overall Officials: Olexiy Kovalyov, Professor, Principal Investigator — Zaporizhzhia State Medical and Pharmaceutical University; Laila Sara Arroyo Mühr, PhD, Study Director — Karolinska Institutet
Locations (1):
- Educational and Scientific Medical Center "Universitetskaya Klinika", Zaporizhzhia State Medical and Pharmaceutical University, Zaporizhzhya, Ukraine

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive health information collected in a conflict-affected setting, and ethical approvals do not permit external sharing of identifiable or de-identified individual-level data.

REFERENCES:
- [Background] Elfstrom M, Gray PG, Dillner J. Cervical cancer screening improvements with self-sampling during the COVID-19 pandemic. Elife. 2023 Dec 12;12:e80905. doi: 10.7554/eLife.80905. PMID 38085566
- [Background] World Health Organization (2022) HPV self-sampling in Sweden leading to faster elimination of cervical cancer. Retrieved from: https://www.who.int/europe/news/item/08-09-2022-hpv-self-sampling-in-sweden-leading-to-faster-elimination-of-cervical-cancer, accessed on 2024-03-05.
- [Background] World Health Organization. (2018). WHO calls for global action on cervical cancer. Retrieved from https://www.who.int/news-room/detail/17-11-2018-who-calls-for-global-action-on-cervical-cancer, accesed on 2024-02-07